CLINICAL TRIAL: NCT02990910
Title: Effects of an Individualized Analgesia Protocol on the Requirements of Medical Interventions After Adenotonsillectomy in Children Based on the Result of a Fentanyl Test: a Randomized Controlled Trial
Brief Title: Individualized Analgesia After Adenotonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xuan Wang, Doctor, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IARA
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Analgesia
Keywords: respiratory adverse events; adenotonsillectomy; opioid analgesia; children
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized opioid analgesia (Other): One group: positive result 10μg/kg morphine; negative result 50μg/kg morphine.Scored every 10 minutes until CHEOPS<=6 and Aldrete score>9.
  Interventions: Drug: Individualized opioid analgesia
- conventional opioid analgesia (Other): Another group: all received 25μg/kg morphine .Scored every 10 minutes until CHEOPS<=6 and Aldrete score>9.
  Interventions: Device: conventional opioid analgesia

INTERVENTIONS:
Drug: Individualized opioid analgesia — (a）positive result 10μg/kg morphine; negative result 50μg/kg morphine.
  Other Names: IP
  Arms: Individualized opioid analgesia
Device: conventional opioid analgesia — (b) all received 25μg/kg morphine
  Other Names: CP
  Arms: conventional opioid analgesia

SUMMARY:
A high incidence of respiratory morbidity after adenotonsillectomy is reported in children with obstructive sleep apnea syndrome (OSAS). So we designed a prospective, double-blind, randomized controlled study to determine the effects of individualized opioid analgesia compared with conventional opioid analgesia on respiratory morbidity after adenotonsillectomy in Children with OSAS.

DETAILED DESCRIPTION:
All children were randomized 2 groups based on a computer-generated random number. The main interventions were occurred in post anesthetic care unit (PACU). In the operating room, all patients received a standardized anesthetic regimen by one anesthetist. Sevoflurane was used for maintenance without any opioids. Before the end of the procedure, spontaneous respiratory was recovered. All the patients were given 1 mcg/kg fentanyl intravenous injection after the end of the procedure. The positive result was defined as spontaneous respiratory rate decreased more than 50%, the others were defined as negative result. The result of fentanyl test submitted to assistant, and prepared the rescue analgesic drugs according to this result. One group: positive result 10μg/kg morphine; negative result 50μg/kg morphine. Another group: all received 25μg/kg morphine .The trachea was extubated when patients were awake, and then transported to the PACU. Patients with a Children's Hospital of Eastern Ontario Pain Scale score>6 received rescue analgesic drugs and observe respiratory morbidity in each group.

ELIGIBILITY:
Inclusion Criteria:

* children with obstructive sleep apnea syndrome undergoing elective T&A, ASA physical status I-II

Exclusion Criteria:

* developmental delay cardiac and craniofacial abnormalities ASA classification III or more body mass index more than the 95th percentile for age

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: xuan wang, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Chilren's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo J, Zhuang P, Liu K, Wan Y, Wang X. Effects of an individualized analgesia protocol on the need for medical interventions after adenotonsillectomy in children: a randomized controlled trial. BMC Anesthesiol. 2021 Feb 8;21(1):41. doi: 10.1186/s12871-021-01263-3. PMID 33557762

RESULTS

PARTICIPANT FLOW:
Recruitment Details: children who scheduled for adenotonsillectomy under general anesthesia
Pre-assignment Details: Patients with a history of allergy, pulmonary or cardiac diseases were excluded.
Groups:
- Individualized Opioid Analgesia: One group: positive result 10μg/kg morphine; negative result 50μg/kg morphine.Scored every 10 minutes until CHEOPS<=6 and Aldrete score>9.
  personalized opioid analgesia: (a）positive result 10μg/kg morphine; negative result 50μg/kg morphine.
Period: Overall Study
Arm/Group | Individualized Opioid Analgesia | Conventional Opioid Analgesia
Started (accorded with the inclusion criteria) | 140 | 140
Completed (back to the wards) | 134 | 130
Not Completed | 6 | 10
Not completed — Lack of Efficacy | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individualized Opioid Analgesia | Conventional Opioid Analgesia | Total
Number analyzed (Participants) | 140 | 140 | 280
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6 [4 to 8] | 5 [4 to 6] | 6 [4 to 8]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The children with cough after intravenous fentanyl, the study was excluded
  Participants
    number analyzed (Participants) | 134 | 130 | 264
    Female | 48 | 52 | 100
    Male | 86 | 78 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 140 | 140 | 280
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 140 | 140 | 280
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 140 | 140 | 280
Region of Enrollment [Number; unit: participants]
  China | 140 | 140 | 280
BMI [Median (Inter-Quartile Range); unit: kg / m^2] | 18 [17 to 20] | 18 [16 to 19] | 18 [16 to 19]

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Requiring at Least One Medical Intervention for Respiratory Events
Description: The medical interventions included instrumentation of the airway, bag/mask ventilation, and/or drug administration (succinylcholine, albuterol, or naloxone), which were classified as major medical interventions. The medical interventions also included repositioning of the child's airway, chin lift/jaw thrust maneuvers, and/or escalating to an oxygen mask, which were classified as minor medical interventions. Since oxygen by nasal cannula was delivered to all children recovering from anesthesia, escalating to an oxygen mask implied the patient need but higher concentration of oxygen to maintain SpO2 ≥ 95%.
Time Frame: Time from entering the PACU until the patient leaves,approx 1 hour.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Opioid Analgesia | Conventional Opioid Analgesia
Number analyzed (Participants) | 134 | 130
Participants | 16 | 29
Statistical Analysis 1: Comparison: Individualized Opioid Analgesia vs Conventional Opioid Analgesia; Chi square test was used to compare the count data,p < 0.05 was considered statistically significant; Test type: Superiority; p < 0.05, Chi-squared

2. Secondary Outcome: The Median Survival Time for CHEOPS Score > 6.
Description: Pain was assessed and recorded through the East Ontario children's hospital pain score (CHEOPS).When the CHEOPS>6,We thought it is painful. Comparing the median survival time (the time corresponding to pain percentage of 50% in two groups) for CHEOPS>6 in two groups.
Time Frame: Time from entering the PACU until the patient leaves,approx 1 hour.
Measure: Median (95% Confidence Interval); unit: minute
Arm/Group | Individualized Opioid Analgesia | Conventional Opioid Analgesia
Number analyzed (Participants) | 134 | 130
minute | 20 [17 to 23] | 30 [28 to 32]

ADVERSE EVENTS:
Time Frame: Time from entering the PACU until the patient leaves,approx 1 hour.
Description: Respiratory adverse events were defined as an intervention requiring a nurse to maintain the SPO2 ≥95%.
Arm/Group | Individualized Opioid Analgesia | Conventional Opioid Analgesia
All-Cause Mortality (participants affected / at risk) | 16/134 | 29/130
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/130
Other Adverse Events (participants affected / at risk) | 16/134 | 22/130
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individualized Opioid Analgesia (N=134) | Conventional Opioid Analgesia (N=130)
Post Operative Nausea And Vomitting (Surgical and medical procedures) | 16 (16) | 22 (22)

LIMITATIONS AND CAVEATS:
The absence of PSG assessment before surgery in patients recruited in this study is a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT02990910/SAP_003.pdf
  • Informed Consent Form (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT02990910/ICF_004.pdf
  • Study Protocol (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT02990910/Prot_005.pdf